CLINICAL TRIAL: NCT05742854
Title: Compariıson Of The Effects Of Carbetocin And Oxytocin, Which Are Uterotonic Agents, In C-Section Operations
Brief Title: Comparison Of The Effects Of Carbetocin And Oxytocin In C-Sectıon
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Asuman Sargın, Principal Investigator, Ege University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ASargın
Record Dates: First submitted 2021-12-28; First posted 2023-02-24 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Carbetocin; Oxytocic Drugs Causing Adverse Effects in Therapeutic Use
Keywords: Carbetocin; C-section; Postpartum hemorrhage; Oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin

STUDY DESIGN:
Intervention Model Description: This study intends to investigate oxytocin and carbetocin, which are uterotonic agents used during C-section, in terms of haemodynamic changes they cause, their effects on the uterine tone and on bleeding as well as their side effects (flushing, headache, back pain, hypertension and tachycardia, nausea-vomiting, etc.), to determine if there are any differences between them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Active Comparator): (subjects administered oxytocin as a uterotonic agent) (5 IU oxytocin diluted with 10 ml saline followed by slow injection) (for 3 minutes)
  Interventions: Procedure: C-sections operations; Drug: Oxytocin
- Carbetocin (Active Comparator): subjects administered carbetocin as a uterotonic agent) (100µg carbetocin diluted with 10 ml saline followed by slow injection (for 3 minutes))
  Interventions: Procedure: C-sections operations; Drug: Carbetocin

INTERVENTIONS:
Procedure: C-sections operations — Immediately after the delivery of the baby, uterotonic agents will be applied before the placenta is removed and by a manual check of the fundus of the uterus and the anterior wall, followed by an examination of the uterine tone by the surgeon
Drug: Oxytocin — Oxytocin
  Arms: Oxytocin
Drug: Carbetocin — Carbetocin
  Arms: Carbetocin

SUMMARY:
Obstetric hemorrhage is the most common cause of maternal mortality worldwide and its incidence is estimated to be approximately 24%. A series of studies has shown that the risk of serious postpartum hemorrhage decreases with correct and active management in the third stage of labor. And the routine use of uterotonic agents underlies effective management. It has been reported that the routine use of uterotonic agents (oxytocin, carbetocin, ergometrine, etc.) reduces the risk of postpartum bleeding by 40% on average. However, the uterotonic agent and dose protocol are still unclear. Oxytocin is the most preferred agent for postpartum hemorrhage prophylaxis after vaginal and cesarean delivery in cases without risk factors, as it has a rapid onset of effect, does not increase blood pressure, and does not cause a retained placenta. In cases where oxytocin cannot be used, other agents of choice are ergot derivatives and misoprostol. The use of carbetocin, a long-acting oxytocin analogue, is now recommended in the guidelines for risky vaginal deliveries and postpartum hemorrhage prophylaxis after C-section. Carbetocin also reduces the need for additional uterotonics. Although carbetocin has been approved for use by the ministry of health, it still has limited clinical use in Turkey. It is vital for the medical community to have more experience with using carbetocin, an agent cited in medical guidelines and is also available in our country, and to share their experiences on academic platforms. This study intends to investigate oxytocin and carbetocin, which are uterotonic agents used during C-section, in terms of haemodynamic changes they cause, their effects on the uterine tone and on bleeding as well as their side effects (flushing, headache, back pain, hypertension and tachycardia, nausea-vomiting, etc.), to determine if there are any differences between them and share our insights with the reader.

DETAILED DESCRIPTION:
Obstetric hemorrhage is the most common cause of maternal mortality worldwide and its incidence is estimated to be approximately 24%. A series of studies has shown that the risk of serious postpartum hemorrhage decreases with correct and active management in the third stage of labor. And the routine use of uterotonic agents underlies effective management. It has been reported that the routine use of uterotonic agents (oxytocin, carbetocin, ergometrine, etc.) reduces the risk of postpartum bleeding by 40% on average. However, the uterotonic agent and dose protocol are still unclear. Oxytocin is the most preferred agent for postpartum hemorrhage prophylaxis after vaginal and cesarean delivery in cases without risk factors, as it has a rapid onset of effect, does not increase blood pressure, and does not cause a retained placenta. In cases where oxytocin cannot be used, other agents of choice are ergot derivatives and misoprostol. The use of carbetocin, a long-acting oxytocin analogue, is now recommended in the guidelines for risky vaginal deliveries and postpartum hemorrhage prophylaxis after C-section. Carbetocin also reduces the need for additional uterotonics. Although carbetocin has been approved for use by the ministry of health, it still has limited clinical use in Turkey. It is vital for the medical community to have more experience with using carbetocin, an agent cited in medical guidelines and is also available in our country, and to share their experiences on academic platforms. This study intends to investigate oxytocin and carbetocin, which are uterotonic agents used during C-section, in terms of haemodynamic changes they cause, their effects on the uterine tone and on bleeding as well as their side effects (flushing, headache, back pain, hypertension and tachycardia, nausea-vomiting, etc.), to determine if there are any differences between them and share our insights with the reader.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Pregnant women to have a C-section,
* Subjects with no history of oxytocin allergy, At term, no multiple pregnancies, elective C-section

Exclusion Criteria:

Subjects refusing to take part,

* Subjects with a history of oxytocin allergy, Subjects scheduled for an emergency C-section, Multiple pregnancies, Having been diagnosed with diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-09 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Effect of uterotonic agents on uterine tone | intraoperative
  uterine tone (standardized as Very good, Good, Sufficient, Atony),
hemorrhage | haemoglobin levels before and after 6 hours.
  haemoglobin concentration

SECONDARY OUTCOMES:
in terms of haemodynamic changes uterotonic agents cause | intraoperative time, after 30 minute
  Blood pressure (in mmHg),hypotansion
side effects of uterotonic agents | postoperative,24 hours after caesarean section
  lushing, headache, back pain, hypertension and tachycardia, nausea-vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- EÜTF, Bornova, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No